CLINICAL TRIAL: NCT02745223
Title: A Phase 2a, Double-blind, Randomized, Placebo-controlled, Repeated Administration, Crossover Study to Establish Safety, Tolerability and Efficacy of PresbiDrops (CSF-1) in Presbyopic Subjects
Brief Title: Safety, Tolerability, and Efficacy of PresbiDrops (CSF-1), a Topical Ophthalmic Drug for Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orasis Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FG-PRE-101
Record Dates: First submitted 2016-03-09; First posted 2016-04-20 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PresbiDrops (CSF-1) (Experimental): Participants self-administered PresbiDrops (CSF-1), 1 drop in each eye each morning for 2 weeks.
  Interventions: Drug: PresbiDrops (CSF-1)
- Placebo (Placebo Comparator): Participants self-administered placebo, 1 drop in each eye each morning for 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PresbiDrops (CSF-1) — PresbiDrops (CSF-1) is a topical ophthalmic drug.
  Arms: PresbiDrops (CSF-1)
Drug: Placebo — Placebo drops contains the same ingredients as PresbiDrops except for the active ingredients.
  Arms: Placebo

SUMMARY:
A study to establish safety, tolerability, and efficacy of PresbiDrops (CSF-1) in presbyopic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 40 and 65 years of age (inclusive).
2. Subjects who provide written informed consent to participate in the study.
3. Subjects have signs of presbyopia upon ophthalmic examination.
4. Subjects have normal presbyopia with low distance refraction (sphere no greater than ±0.75 diopter cylinder no greater than ±0.75 diopter cylinder [DC], refraction along any principal meridian no greater than 1.00 diopter).
5. Subjects must have best corrected vision of 20/20 in both eyes, and currently depend on reading glasses or bifocals in which the near addition is > +1.00 diopter.
6. Subjects in general good health in the opinion of the Investigator as determined by medical history.
7. Women with childbearing potential must have a negative urine pregnancy test at Screening and be willing and able to use a medically acceptable method of birth control or they must be postmenopausal. Acceptable methods of birth control in this study include: Vasectomy, tubal ligation, consistent use of an approved oral contraceptive (birth control pill), intrauterine device (IUD), hormonal implants, contraceptive injection or a double barrier method (diaphragm with spermicidal gel or condom with contraceptive foam). Postmenopausal women are defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.
8. Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study.

Exclusion Criteria:

1. History of macular disease or any other ocular conditions or congenital malformation.
2. Any medical condition known to affect the structure of the uvea, cornea, lens, or retina or main function of the eyes.
3. No cataract or minimal nuclear sclerosis.
4. Severe dry eye.
5. Any topical ophthalmic medications, other than artificial tears (up to a maximum of 4 times per day) and medications that are associated with fluctuation of accommodative capacity and/or pupil size, unless on a stable dose for at least 3 months before the Screening visit.
6. Contact lenses for the past three months before the Screening visit.
7. A difference of more than 0.50 diopter between the manifest spherical equivalent and the wave front refraction spherical equivalent.
8. Pupil size less than 2,5 mm in either eye prior to dilation at ambient light of 8-15 lux prior to the Baseline visit.
9. A history of herpes (of any kind) in either eye.
10. Cataract surgery and/or refractive surgery in either eye.
11. Known contraindication, hypersensitivity, and/or allergy to any study drugs or excipients.
12. Any acute illness (eg, acute infection) within 48 hours of first study drug administration, which is considered of significance by the Investigator.
13. Participation in another clinical trial with drugs received within 30 days of Screening.
14. Pregnant or currently lactating women.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a ≥ 2 line improvement from Baseline in uncorrected near distance visual acuity | Baseline to end of treatment (up to 14 days)
  Uncorrected visual acuity will be assessed at distance and near (40 cm) using a standardized eye chart. The number of lines in the eye chart that the participant correctly identifies will be measured. The test will be performed both binocularly and on 1 eye at a time by covering the eye not being tested. Distance visual acuity will be measured under normal light conditions. Near acuity will be measured both in poor light conditions and normal light conditions.
Mean change from Baseline in the number of lines correctly identified in uncorrected near distance visual acuity | Baseline to end of treatment (up to 14 days)
  Uncorrected visual acuity will be assessed at distance and near (40 cm) using a standardized eye chart. The number of lines in the eye chart that the participant correctly identifies will be measured. The test will be performed both binocularly and on 1 eye at a time by covering the eye not being tested. Distance visual acuity will be measured under normal light conditions. Near acuity will be measured both in poor light conditions.

SECONDARY OUTCOMES:
Percentage of participants with a ≥ 2 line improvement from Baseline in uncorrected intermediate distance visual acuity | Baseline to end of treatment (up to 14 days)
  Uncorrected visual acuity will be assessed at distance and intermediate (60 cm) using a standardized eye chart. The number of lines in the eye chart that the participant correctly identifies will be measured. The test will be performed both binocularly and on 1 eye at a time by covering the eye not being tested. Distance and intermediate visual acuity will be measured under normal light conditions.
Mean change from Baseline in the number of lines correctly identified in uncorrected intermediate distance visual acuity | Baseline to end of treatment (up to 14 days)
  Uncorrected visual acuity will be assessed at distance and intermediate (60 cm) using a standardized eye chart. The number of lines in the eye chart that the participant correctly identifies will be measured. The test will be performed both binocularly and on 1 eye at a time by covering the eye not being tested. Distance and intermediate visual acuity will be measured under normal light conditions.
Change from Baseline in the depth of focus at distance and near | Baseline to end of treatment (up to 14 days)
  Depth of focus (DoF) is defined as the distance in diopters that a viewed object can be moved towards or away from the eye until the object is no longer judged to be in focus. DoF will be assessed using either wavefront aberrometry or according to the following instructions. Distance: Set the distance spectacle prescription in the refractor head/trial frame. Have the participant look at the 6/9 (0.6) Snellen letter. Increase the plus sphere power until the participant reports blurring (+a diopters). Repeat using negative lenses (-b diopters). Remove the negative sign in front of b. Depth of focus at distance = (a+b) diopters. Near: Set the distance spectacle prescription at +2.5 diopters in the refractor head/trial frame. Have the participant look at the J2 print at 40 cm. Increase the plus sphere power until the participant reports blurring (+x diopters). Repeat using negative lenses (-y diopters). Remove the negative sign in front of y. The depth of focus at near = (x+y) diopters.
Change from Baseline in uncorrected distance visual acuity | Baseline to end of treatment (up to 14 days)
  Uncorrected visual acuity will be assessed at distance using a standardized eye chart under normal light conditions. The test will be performed both binocularly and on 1 eye at a time by covering the eye not being tested.
Change from Baseline in the need for glasses | Baseline to end of treatment (up to 14 days)
  The Patient Reported Outcome Questionnaire includes 29 questions assessing subject satisfaction of their vision and the need for eye glasses in order to perform daily tasks.
Change from Baseline in pupil diameter and appearance | Baseline to end of treatment (up to 14 days)
  Pupil size and appearance will be evaluated by wave-front aberrometer. Examination will be conducted at near mesopic conditions, in low but not quite dark lighting situations at a fixed setting on the light meter. Mesopic light levels range from luminance of approximately 0.001 to 3 cd m-2, an appropriate and fixed setting will be selected, that reflects most night-time outdoor and traffic lighting scenarios. An examination of pupillary function includes inspecting the pupils for equal size (1 mm or less of difference may be normal), regular shape, reactivity to light, and direct and consensual accommodation (PERRLA [D+C]; Pupils Equal and Round, Reactive to Light and Accommodation [Direct and Consensual]).
Change from Baseline in the stability of pre-corneal tear film | Baseline to end of treatment (up to 14 days)
  Assessment of the stability of pre-corneal tear film will be conducted using non-invasive break up time (NIBUT) and tear meniscus height. NIBUT is measured with instruments such as a Keratometer, a hand-held Keratoscope, or a Tearscope. After a blink, the reflection observed with these instruments is clear and crisp when the ocular surface is free from any irregularities. NIBUT is defined as the interval between the opening of the eyes and the moment when an irregularity is observed. NIBUT values < 10 seconds indicate dry eyes. Tear meniscus height (TMH) can be measured with a slit-lamp biomicroscope. A slit lamp image of the lower TMH can be photographed or captured electronically and later measured directly on screen and corrected for magnification. The lower TMH represents the total volume of tears at the ocular surface. Heights of less than 0.2 mm indicate reduced tear volume. A tear meniscus with a scalloped edge is often associated with a dry eye.
Change from Baseline in visual field | Baseline to end of treatment (up to 14 days)
  Testing the visual fields will consist of confrontation field testing in which each eye is tested separately to assess the extent of the peripheral field. Visual field is assessed in each eye separately. The participant occludes 1 eye while fixated on the examiner's eye with the non-occluded eye. The subject is then asked to count the number of fingers that are briefly flashed in each of 4 quadrants (left, right, up, and down).

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Blumental, Study Director — Head of Ophthalmology Department, Rambam Medical Center, Haifa, Israel; Andreja Veselica, Study Director — VID Medical Center, Nova Gorica, Slovenia
Locations (1):
- The Department of Ophthalmology, Rambam Health Care Campus, Haifa, Israel